CLINICAL TRIAL: NCT00562510
Title: A Phase 3, Randomized, Double Blinded, Placebo Controlled Study of Raltegravir Added to Stable HAART in HIV-1 Infected Subjects With Viral Suppression and Low CD4 Recovery
Brief Title: Raltegravir Added to Stable HAART in HIV-1 Infected Subjects With Viral Suppression and Low CD4 Recovery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment lower than estimated
Sponsor: Pedro Cahn (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Pedro Cahn, MD, Fundación Huésped
Organization: Fundación Huésped (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FH-RAL-01; ANMAT-1-4721846/07-6
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; raltegravir; immune discordance; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir
- Raltegravir matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg BID added to stable HAART
  Arms: Raltegravir
Drug: Placebo — Placebo BID added to stable HAART
  Arms: Raltegravir matching placebo

SUMMARY:
This is a Phase 3, randomized, double blinded, placebo-controlled study designed to compare the safety, tolerability, antiviral activity and immunological effect of raltegravir added to a previously stable HAART regimen in the treatment of HIV-1 infected subjects with undetectable viraemia and low CD4 recovery.

HYPOTHESIS:

Adding raltegravir to a stable HAART in patients with undetectable plasma viral load and low CD4 recovery will result in further viral suppression and therefore higher CD4 recovery.

DETAILED DESCRIPTION:
Although HAART has reduced the morbidity and mortality from HIV-1 infection, some patients experience a discordant response characterized by HIV-1 RNA plasma levels below the limit of detection and low CD4 T-cell recovery (immunologic discordant responders). At present, recommendations for the clinical management of patients with discordant responses to antiretroviral therapy are largely based on observational, uncontrolled data.

The effect on CD4 count of adding raltegravir in already undetectable patients has not yet been evaluated.

The primary purpose of this study is to assess the ability of the HIV-1 integrase inhibitor, raltegravir, added to a stable HAART, to increase CD4 count in patients with undetectable plasma viral load and low CD4 recovery.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Subject has voluntarily signed and dated an informed consent form.
* Documented sustained HIV RNA < 50 copies/ml (two consecutive pVL < 50 copies/ml, first VL > 12 months before the screening date) without documentation of HIV RNA > 50 copies/ml for at least 12 months while on previous stable HAART (PS_HAART).
* HIV RNA < 50 copies/ml at screening.
* Subject is currently receiving an antiretroviral regimen which has not changed for at least 12 months.
* CD4 count < 200 cells/ mm3 AND CD4 increase < 100 cells/ mm3 in the last 12 months.
* Subject's vital signs, physical examination and laboratory results do not exhibit evidence of acute illness.
* Negative serum or urine pregnancy test and willing to use acceptable means of contraception.

Exclusion Criteria:

* Patient is receiving tenofovir DF AND didanosine as a component of the background antiretroviral therapy.
* Patient has a current (active) diagnosis of acute hepatitis due to any cause OR chronic hepatitis B and/or C WITH aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>2.5 x upper limit of normal (ULN) AND/OR is likely to require treatment in the next year.
* Subject has significant history of cardiac, renal, neurologic, psychiatric, oncologic, metabolic, or hepatic disease or any condition that, in the investigators opinion, could compromise the subject's safety or adherence to the trial protocol.
* Subject has a currently active AIDS defining illness (category C conditions according to the CDC Classification System for HIV infection 1993) within 30 days of screening. Subjects who are on stable maintenance therapy for an opportunistic infection may be enrolled.
* Life expectancy < 1 year according to the judgment of the investigator.
* Screening laboratory analysis show any of the following abnormal laboratory results:

  * Hemoglobin < 8.0 g/dL
  * Absolute neutrophil count < 750 cells/µL
  * Platelet count < 50,000 mm3
* Use of any investigational agents within 30 days prior to screening.
* Previous use of integrase inhibitors.
* Use of immunosuppressive drugs, cytokine inhibitors or other cytokines in the last year.
* Continuous use of systemic corticoids for more than a month in the last year or any use in the last 3 months.
* Subject has an ongoing history of substance abuse or psychiatric illness.
* Subject is pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects increasing CD4 count > 50 cells/mm³. | 48 weeks

SECONDARY OUTCOMES:
Proportion of patients achieving plasma HIV-RNA < 5 copies/ml. | 48 weeks
Proportion of subjects increasing CD4 count > 50 cells/mm³. | 24 weeks
Proportion of patients achieving CD4 count > 250 cells/mm3 | 48 weeks
Proportion of patients achieving an increase of 5 percentual points in CD4 percentage | 48 weeks
Median change from baseline in CD4 count. | 48 weeks
Proportion of patients maintaining HIV RNA <50 copies/ml. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Cahn, MD, PhD, Principal Investigator — Fundacion Huesped
Locations (1):
- Fundacion Huesped, Buenos Aires, Argentina

REFERENCES:
- See also: Fundacion Huesped — http://www.huesped.org.ar